CLINICAL TRIAL: NCT00398112
Title: A Phase II Study of Sunitinib Malate for Treatment of Patients With Relapsed/Refractory Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL)
Brief Title: Sunitinib in Treating Patients With Relapsed or Refractory Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01830; NCI-2012-01830 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCCTG-N0683; CDR0000512979; N0683 (Other: North Central Cancer Treatment Group); N0683 (Other: CTEP); U10CA025224 (NIH)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2012-12

CONDITIONS: B-cell Chronic Lymphocytic Leukemia; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Sunitinib

ARMS (1):
- Arm I (Experimental): Patients receive oral sunitinib malate daily on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sunitinib malate; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sunitinib malate — Given orally
  Other Names: SU11248; sunitinib; Sutent
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well sunitinib works in treating patients with relapsed or refractory chronic lymphocytic leukemia or small lymphocytic lymphoma. Sunitinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the response rate (complete response [CR] and partial response) in patients with relapsed or refractory chronic lymphocytic leukemia or small lymphocytic lymphoma treated with sunitinib malate.

II. Assess the toxicity of this drug in these patients. III. Assess duration of response, time to progression, overall survival, and CR rate in patients treated with this drug.

SECONDARY OBJECTIVES:

I. Evaluate if known risk stratification parameters (i.e., immunoglobulin mutational status, ZAP-70 status, fluorescent in situ hybridization [FISH] defects, and/or CD38 status) are related to clinical response to sunitinib malate.

OUTLINE: This is a multicenter study.

Patients receive oral sunitinib malate daily on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

Patients undergo blood collection periodically for translational and pharmacological studies, including IgVH gene mutation status and ZAP-70 status. Samples are examined by fluorescent in situ hybridization (FISH) and other assays.

After completion of study treatment, patients are followed every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of 1 of the following:

  * Biopsy proven small lymphocytic lymphoma (SLL)
  * Chronic lymphocytic leukemia (CLL) meeting all of the following criteria:

    * Peripheral blood lymphocyte count > 5,000/mm^3
    * Lymphocytes must consist of small to moderate size lymphocytes, with < 55% prolymphocytes, atypical lymphocytes, or lymphoblasts morphologically
    * Immunophenotyping consistent with CLL, defined by the following criteria:

      * Predominant population of lymphocytes share both B-cell antigens (i.e., CD19, CD20, or CD23) as well as CD5 in the absence of other pan-T-cell markers (e.g., CD3 or CD2)
      * Dim surface immunoglobulin expression
      * Exclusively kappa and lambda light chains
      * Splenomegaly, hepatomegaly, or lymphadenopathy are not required
* Refractory or relapsed disease as evidenced by 1 of the following criteria:

  * Progression after ≥ 1 course of a purine nucleoside (i.e., fludarabine phosphate, cladribine, pentostatin) regimen
  * Progression after ≥ 1 course of an alkylator (i.e., cyclophosphamide or chlorambucil) regimen
  * Relapse after ≥ 1 prior purine nucleoside oral kylator (i.e., cyclophosphamide or chlorambucil) regimen
* Requires chemotherapy, as indicated by any of the following criteria:

  * Measurable (i.e., > 5,000/mm^3) and progressive clonal lymphocytosis
  * Measurable (i.e., single diameter > 2 cm) and progressive lymphadenopathy
  * Disease-related symptoms, including 1 or more of the following:

    * Weight loss > 10% within the past 6 months
    * Extreme fatigue attributed to CLL/SLL
    * Fevers > 100.5^oF for 2 weeks without evidence of infection
    * Night sweats without evidence of infection
  * Evidence of progressive marrow failure, as manifested by the development of or worsening anemia (hemoglobin < 10 g/dL) and/or thrombocytopenia (platelet count < 100,000/mm^3)
  * Massive (i.e. > 6 cm below left costal margin) or progressives plenomegaly
* No mantle cell lymphoma, as demonstrated by a negative fluorescent in situ hybridization (FISH) analysis fort(11;14)(IgVH/CCND1) on peripheral blood or tissue biopsy
* ECOG performance status 0-2
* Life expectancy ≥ 12 months
* Creatinine ≤ 1.5 times upper limit of normal (ULN) OR creatinine clearance ≥ 60 mL/min
* AST and ALT ≤ 2.5 times ULN
* Bilirubin normal
* Alkaline phosphatase ≤ 3 times ULN
* Platelet count > 30,000/mm^3 (without transfusion)
* Absolute neutrophil count > 1,000/mm^3
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to complete patient diaries alone or with assistance
* No abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 28 days
* No other malignancy except for squamous cell or basal cell carcinoma of the skin or in situ carcinoma of the cervix, unless the tumor was curatively treated within the past 2 years
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to sunitinib malate
* No inability to swallow or retain sunitinib malate capsules due to any of the following:

  * Gastrointestinal tract disease
  * Requirement for IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* No pre-existing thyroid abnormality that would make the patient unable to maintain normal thyroid function with medication
* No pulmonary embolism within the past 12 months
* No serious or nonhealing wound, ulcer, or bone fracture
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infections
  * Psychiatric illness or social situation that would limit compliance with study requirements
* No cerebrovascular accident or transient ischemic attack within the past 12 months
* No uncontrolled hypertension (i.e., systolic blood pressure [BP] ≥ 140 mm Hg or diastolic BP ≥ 90 mm Hg)
* No significant cardiac arrhythmia, including any of the following:

  * QTc prolongation (i.e., QTc interval ≥ 500 msec)
  * Ventricular tachycardia
  * Atrial fibrillation
  * Atrial flutter
  * Second or third degree heart block
* No cardiac disease within the past 12 months, including any of the following:

  * Myocardial infarction
  * Cardiac arrhythmia
  * Stable/unstable angina
  * Symptomatic congestive heart failure
  * Coronary/peripheral artery bypass graft or stenting
* No New York Heart Association (NYHA) class III or IV heart failure

  * The following patients are eligible provided they have NYHA class II cardiac function on baseline ECHO/MUGA:

    * History of NYHA class II heart failure and asymptomatic on treatment
    * No prior anthracycline exposure
    * No prior central thoracic radiation that included the heart in the radiation port
* See Disease Characteristics
* At least 4 weeks since prior chemotherapy
* At least 4 weeks since prior rituximab or alemtuzumab
* At least 4 weeks since prior major surgery
* At least 4 weeks since prior oral steroids
* No prior treatment with any other antiangiogenic agent, including any of the following:

  * Bevacizumab
  * Sorafenib
  * Pazopanib
  * AZD2171
  * Vatalanib
  * VEGF Trap
* At least 7 days since prior and no concurrent CYP3A4 inhibitors, including any of the following:

  * Ketoconazole
  * Itraconazole
  * Clarithromycin
  * Erythromycin
  * Diltiazem
  * Verapamil
  * HIV protease inhibitors (i.e., indinavir, saquinavir,ritonavir, atazanavir, nelfinavir)
  * Delavirdine
* At least 12 days since prior and no concurrent CYP3A4 inducers, including any of the following:

  * Rifampin
  * Rifabutin
  * Carbamazepine
  * Phenobarbital
  * Phenytoin
  * Hypericum perforatum (St. John's wort)
  * Efavirenz
  * Tipranavir
* No other concurrent investigational agents
* No concurrent agents with proarrhythmic potential, including any of the following:

  * Terfenadine
  * Quinidine
  * Procainamide
  * Disopyramide
  * Sotalol
  * Probucol
  * Bepridil
  * Haloperidol
  * Risperidone
  * Indapamide
  * Flecainide
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer agents or therapies
* No concurrent therapeutic doses of coumarin-derivative anticoagulants (e.g., warfarin)

  * Concurrent prophylactic low molecular weight heparin or warfarin at doses ≤ 2 mg daily for thrombosis prophylaxis allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-08; Primary Completion 2008-11 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tait Shanafelt, Principal Investigator — North Central Cancer Treatment Group
Locations (1):
- North Central Cancer Treatment Group, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between August 2007 and December 2008, 18 participants were recruited.
Pre-assignment Details: All participants were eligible and included in all analyses.
Groups:
- Sunitinib Malate: Patients receive oral sunitinib malate 37.5 mg daily on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Sunitinib Malate
Started | 18
Completed | 0
Not Completed | 18
Not completed — Adverse Event | 4
Not completed — Disease progression | 9
Not completed — Alternative treatment | 1
Not completed — Withdrawal by Subject | 3
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 18
Age, Continuous [Median (Full Range); unit: years] | 67.5 [51 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 18
Fluorescence In Situ Hybridization (FISH) Abnormalities [Number; unit: participants] — FISH abnormalities were categorized according to Dohner hierarchy. This test determines the presence of abnormalities in specific chromosomes of CLL cells, which are associated with more or less aggressive forms of cancer. Patients with abnormalities of chromosome 11 (deletion 11q23) and 17 (deletion 17p13) experience rapid progression of their CLL.
  participants
    del 17p13 | 6
    del 11q23 | 1
    Trisomy 12 | 5
    del 13q14 | 2
    Normal | 4
Rai Stage [Number; unit: participants] — Rai staging is a way to categorize the disease progression of chronic lymphocytic leukemia (CLL); higher stages reflect increasing severity.
  Rai Stage 0: Lymphocytosis only; Rai Stage I: Lymphocytosis and lymphadenopathy; Rai Stage II: Lymphocytosis and hepatomegaly +/- splenomegaly; Rai Stage III: Lymphocytosis and anemia; Rai Stage IV: Lymphocytosis and thrombocytopenia
  participants
    Low (Rai 0) | 0
    Intermediate (Rai I-II) | 8
    High (Rai III-IV) | 10
ZAP-70 Status [Number; unit: participants] — This test is used to predict the rate of progression from diagnosis to need for treatment in CLL. Participants with positive ZAP-70 (>=20%) tend to experience a more aggressive course of CLL.
  participants
    Positive | 10
    Negative | 8
CD38 Status [Number; unit: participants] — This test is used to predict the rate of progression from diagnosis to need for treatment in CLL. Participants with positive CD38 (>=30%) tend to experience a more aggressive course of CLL.
  participants
    Positive | 9
    Negative | 9
Immunoglobulin Variable Heavy Chain (IGVH) Mutation Status [Number; unit: participants] — IGVH testing helps predict which patients will experience a more aggressive (if the gene is unmutated, <=2%) or less aggressive (if the gene is mutated, >2%) course of CLL. This technically complex test is only available at select medical institutions.
  participants
    Unmutated | 1
    Mutated | 0
    Missing | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Confirmed Response [Complete Response (CR) and Partial Response (PR)] on 2 Consecutive Evaluations at Least 4 Weeks Apart
Description: National Cancer Institute working group criteria (NCIWG) was used to assess response.>
  * CR: no lymphadenopathy, hepatomegaly, splenomegaly or constitutional symptoms; normal complete blood count; confirmed by bone marrow (BM) aspirate & biopsy>
  * PR: 50% decrease in peripheral blood lymphocytes, lymphadenopathy, liver/spleen size, presence/absence of constitutional symptoms; plus ≥1 of the following: ≥1500/μL polymorphonuclear leukocytes, >100000/μL platelets, >11.0 g/dL hemoglobin or 50% improvement for these parameters without transfusions
Time Frame: Duration of Treatment (up to 12 cycles)
Measure: Number; unit: participants
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 18
participants | 0

2. Secondary Outcome: Complete Response Rate in Patients With B-cell Chronic Lymphocytic Leukemia
Description: Complete response is described in the primary outcome
Time Frame: Duration of Treatment (up to 12 cycles)
Population: No participants had a confirmed response, there for this analysis cannot be completed.
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 0

3. Secondary Outcome: Survival Time
Description: Survival time was defined as the time from registration to death due to any cause. The distribution of survival time was estimated using the Kaplan-Meier method.
Time Frame: Duration of study (up to 2 years)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 18
Months | 20.6 [8.0 to NA] — The upper limit of 95% confidence interval of median survival time has not been attained because of the insufficient number of participants with events.

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from registration to progression or death due to any cause. The distribution of PFS was estimated using the Kaplan-Meier method.
Time Frame: Duration of study (up to 2 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 18
months | 2.7 [1.8 to 4.6]

5. Secondary Outcome: Duration of Response
Description: Duration of response was calculated from the documentation (date) of first response (CR or PR) until the date of progression or last follow-up in the subset of patients who responded. The median duration of response with 95%CI was estimated using the Kaplan Meier method
Time Frame: Duration on study (up 2 years)
Population: No participants had a confirmed response, there for this analysis cannot be completed.
Arm/Group | Sunitinib Malate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Sunitinib Malate
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 18/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sunitinib Malate (N=18)
Hemoglobin decreased (Blood and lymphatic system disorders) | 15 (27)
Vision blurred (Eye disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (9)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (7)
Anal mucositis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (11)
Diarrhea (Gastrointestinal disorders) | 8 (18)
Dry mouth (Gastrointestinal disorders) | 2 (9)
Dyspepsia (Gastrointestinal disorders) | 5 (10)
Esophageal mucositis (Gastrointestinal disorders) | 5 (11)
Gastric mucositis (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 10 (16)
Nausea (Gastrointestinal disorders) | 7 (14)
Vomiting (Gastrointestinal disorders) | 3 (6)
Chest pain (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 16 (40)
Localized edema (General disorders) | 2 (5)
Anal infection (Infections and infestations) | 1 (1)
Anorectal infection (Infections and infestations) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (2)
Infectious colitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3)
Alkaline phosphatase increased (Investigations) | 6 (9)
Aspartate aminotransferase increased (Investigations) | 7 (12)
Bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 4 (5)
Leukocyte count decreased (Investigations) | 1 (1)
Lipase increased (Investigations) | 4 (4)
Neutrophil count decreased (Investigations) | 10 (25)
Platelet count decreased (Investigations) | 17 (34)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 10 (19)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 4 (5)
Serum potassium increased (Metabolism and nutrition disorders) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 2 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (5)
Taste alteration (Nervous system disorders) | 4 (9)
Anxiety (Psychiatric disorders) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (9)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2 (3)
Rash desquamating (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertension (Vascular disorders) | 5 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less